CLINICAL TRIAL: NCT00470808
Title: The Effect of a Natural Polyphenolic Extract From Pomegrnate (POMX) on the Development of Atherosclerosis in Diabetic Patients
Acronym: POMX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0051-07-EMC
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-04

CONDITIONS: Atherosclerosis
Keywords: Minors; Enrollment in another study; Males; HBA1C greater than 7; Drug therapy for DM
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: POMx

SUMMARY:
Diabetes is a highly atherogenic disease. Pomegranate juice has impressive antioxidant properties. It has been proven to decrease oxidant stress and to cause the regression of atherosclerotic plaques in hypercholestrolemic and diabetic patients.Furthermore it has been proven to potentiate the biologic activity of the enzyme paraoxonase 1 which is very important in preventing atherosclerosis. The study will try to prove that a polyphenolic extract from pomegranate (POMx) has the same desired effects.

ELIGIBILITY:
Inclusion Criteria:

* Males
* HBA1C>7%
* Drug therapy given for DM

Exclusion Criteria:

* Age<18
* Inclusion in another study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wasseem Rock, MD, Principal Investigator — Ha'Emek Medical Center
Locations (1):
- Ha'Emek Medical Center, Afula, Israel